CLINICAL TRIAL: NCT03335059
Title: A Multicenter, Single-Arm Study Evaluating the Efficacy of Synergo® Radiofrequency-Induced Thermochemotherapy Effect (RITE) With Mitomycin C (Synergo® RITE + MMC) in CIS Non-Muscle Invasive Bladder Cancer (NMIBC) Bacillus Calmette-Guérin (BCG)-Unresponsive Patients With or Without Papillary NMIBC
Brief Title: Mitomycin C Intravesical Chemotherapy in Conjunction With Synergo® Radiofrequency-Induced Hyperthermia for Treatment of Carcinoma in Situ Non-Muscle Invasive Bladder Cancer Patients Unresponsive to Bacillus Calmette-Guérin, With or Without Papillary Tumors.
Acronym: RITE-USA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: poor enrollment
Sponsor: Medical Enterprises Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RITE-1
Record Dates: First submitted 2017-10-30; First posted 2017-11-07 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Bladder Cancer; Bladder Neoplasm; Bladder Tumors; Cancer of Bladder; Cancer of the Bladder; Malignant Tumor of Urinary Bladder; Neoplasms, Bladder; Urinary Bladder Cancer; Carcinoma in Situ of Bladder; Papillary Carcinoma of Bladder (Diagnosis); BCG-Unresponsive Bladder Cancer
Keywords: BCG; Bacillus Calmette-Guérin; CIS; BCG-unresponsive; Synergo; chemohyperthermia; thermochemotherapy; RF; radio frequency; RITE
MeSH Terms: conditions — Urinary Bladder Neoplasms; Disease | interventions — Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Synergo® RITE + MMC (Experimental): Bladder radiofrequency-induced hyperthermia will be delivered in combination with each instillation of MMC in accordance with the Sponsor operational guidelines.
  Interventions: Combination Product: Synergo® RITE + MMC

INTERVENTIONS:
Combination Product: Synergo® RITE + MMC — Subjects will receive a series of induction followed by a series of maintenance bladder instillations of Synergo® RITE + MMC
  Other Names: radiofrequency hyperthermia with mitomycin C; RF hyperthermia with mitomycin C; thermochemotherapy; chemohyperthermia; CHT; radio-frequency hyperthermia with mitomycin C

SUMMARY:
This study will determine whether Synergo® RITE + MMC treatment is efficacious as second-line therapy for CIS NMIBC BCG-unresponsive patients with or without papillary NMIBC, through examination of the complete response rate (CRR) and disease-free duration for complete responders. The study will also explore progression-free survival time, bladder preservation rate, and overall survival time.

The study will address an unmet need to identify a treatment effective in both ablating the disease and providing a prolonged disease-free period for patients. Ideally, the treatment will delay progression to invasive disease, thus preserving the bladder.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with current CIS of the bladder, with or without coexisting papillary Ta/T1 NMIBC tumor(s), who experienced an occurrence or recurrence of CIS within 12 months of completion of adequate BCG7 therapy. An adequate BCG regimen shall consist of at least 2 courses of BCG where the first course (induction) must have included at least 5 of 6 weekly treatments and the second course may have included a re-induction (at least 2 of 6 treatments) or maintenance, (at least 2 of 3 treatments) administered on a schedule similar to the SWOG 8507 study regimen.
2. All clinical, intra-operative and pathological items for the AUA risk stratification must be documented. This includes bladder mapping, according to the instructions specified in the protocol. With regard to BCG and/or other NMIBC treatments documentation must include:

   1. Date of initial treatment,
   2. Date of last treatment,
   3. The number of courses administered and the number of treatments administered in each course.
3. Patients with concomitant papillary tumor(s) must have undergone a repeat TUR 2-4 weeks prior to the first study treatment:

   1. if the previous TUR was incomplete,
   2. if there was no muscle in the specimen after the initial TUR (except in TaLG tumors),
   3. in all T1,
   4. in all HG tumors ≥ 3cm.
4. CT-IVU or MRI-IVU or IVU/retrograde confirmation of absence of tumor(s) in the upper tract, kidney and ureters performed within 6 months before the study treatment initiation, in selected cases, as recommended in latest AUA guidelines published prior to screening. If IVU/retrograde protocol is not available or contrast allergy/poor renal function preclude such imaging, then non-contrast CT or MRI of the abdomen/pelvis within the same timeframe will suffice.
5. Visual inspection to exclude urothelial carcinoma (UC) in the urethra during cystoscopy.
6. Biopsy of the prostatic urethra, prior to enrollment, to exclude UC of the prostatic urethra, in male patients with:

   1. tumor of trigone,
   2. tumor of bladder neck, or
   3. abnormal prostatic urethra
   4. prior history of prostatic urethral involvement.
7. All patients must have urine cytology collected from either voided urine or bladder wash within the screening period prior to enrollment. Patients with positive cytology must also have selective cytology from the upper tract and prostatic urethral biopsies collected within the same period. Patients with a localizing positive upper tract cytology are excluded from the study until definitive treatment renders them free of disease visually and/or radiographically and cytologically (nephroureterectomy, distal ureterectomy or upper tract therapy).
8. Age ≥ 18 yrs.
9. No evidence of urothelial cancer in either kidneys or ureters.
10. Pre-treatment hematology and biochemistry values within the limits:

    1. Hemoglobin ≥ 10 g/dl (g/100 ml)
    2. Platelets ≥ 150 x 10^9/L (x 10^3/mm^3)
    3. WBC ≥ 3.0 x 10^9/L (x 10^3/mm^3)
    4. ANC ≥ 1.5 x 10^9/L (x 10^3/mm^3)
    5. Serum creatinine < 2 mg/dl
    6. SGOT < 1.5 x ULN
    7. SGPT < 1.5 x ULN
    8. Alkaline phosphatase < 1.5 x ULN
11. Negative pregnancy test for women of childbearing potential.
12. A life expectancy at least of the duration of the study.
13. Signed informed consent.

Exclusion Criteria:

1. Non-UC tumor of the urinary tract.
2. Upper tract and/or intramural tumors (e.g., in ostium).
3. Positive selective cytology from the upper tract.
4. History of stage > T1 UC.
5. Papillary tumors > T1 in repeat TUR.
6. Known or suspected reduced bladder capacity. Patients will have an ultrasonic estimation of maximum bladder capacity or void spontaneously the maximum they can retain in their bladder, and this will be used to determine urine volume. A minimum volume of 250 ml is required.
7. Patients with severe bladder outlet obstruction not adequately controlled with medication (AUA symptom score ≥ 20).
8. Bleeding disorder.
9. Gross hematuria within the past 2 weeks before treatment start.
10. Lactating women.
11. Women of childbearing potential unwilling or unable to use adequate contraception if sexually active.
12. More than low-dose methotrexate (>17.5 mg once a week).
13. Other malignancy within the past 5 years, except: non melanomatous skin cancer cured by excision, surgically treated carcinoma in situ of the cervix or ductal CIS (DCIS)/lobular CIS (LCIS) of the breast or stable prostate cancer (under active surveillance or hormone control) with a life expectancy of more than 5 years.
14. Any known allergy (e.g., to MMC) or adverse event that would prevent a prospective study participant from receiving the study treatment.
15. Known untreated urethral strictural disease or bladder neck contracture or any other condition that may prevent catheterization with a 21F catheter. Patients may undergo dilation or urethral incision before entering the study.
16. Bladder diverticulum with diameter > 1cm, as determined by CT or cystography
17. UTI at any time within 3 weeks before study treatment initiation.
18. Significant urinary incontinence (spontaneous, requiring use of > 1 pad/day (PPD)).
19. History of pelvic irradiation.
20. Patients with electronic devices implanted in abdominal cavity.
21. Participation in another study, unless discussed with and approved by the Sponsor or Sponsor's authorized representative.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-02-26 (Actual)

PRIMARY OUTCOMES:
complete response rate (CRR) | 3 months after the initiation of study therapy
  * no CIS
  * no papillary HG tumor
  * no papillary T1 tumor
  * no extra-vesical UC tumor
  * no progression
  a patient will be considered a complete responder only if all the criteria above are met.
  Patients experiencing a new occurrence of a benign tumor or low-grade Ta will be allowed to continue in the study (tumor will be resected); such an occurrence will not constitute an event in the primary analysis.
  Patients with tumors of the ostium and/or upper tract and/or prostatic urethra will be considered to have achieved a complete response in the primary analysis but will be removed from the study.

SECONDARY OUTCOMES:
disease-free duration of complete response (DCR) | through study completion, up to 33 months
  time of recurrence for complete response patients from the 3-month visit until the time of recurrence or until the last follow-up, whichever occurs sooner.

CONTACTS AND LOCATIONS:
Overall Officials: Michael A O'Donnell, MD, Principal Investigator — University of Iowa
Locations (4):
- United States (4):
  - Chesapeake Urology Research Associates, Hanover, Maryland
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No